CLINICAL TRIAL: NCT03878108
Title: Effect of Low Fat Versus Low Carbohydrate Diets on Energy Metabolism
Brief Title: Effects of Low Fat Versus Low Carbohydrate Diets on Energy Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 190067; 19-DK-0067 (Other: NIH Clinical Center)
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Results first posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2020-12-04

CONDITIONS: Healthy; Healthy Volunteers
Keywords: Accelerometry; Body Composition; Body Weight Regulation; Calories; Energy Expenditure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LCHF diet then LFHC diet (Active Comparator): Low carbohydrate, high fat (LCHF) diet then low fat, high carbohydrate diet (LFHC) diet
  Interventions: Dietary Supplement: LCHF diet; Dietary Supplement: LFHC diet
- LFHC diet then LCHF diet (Active Comparator): Low fat, high carbohydrate diet (LFHC) diet then low carbohydrate, high fat (LCHF) diet
  Interventions: Dietary Supplement: LCHF diet; Dietary Supplement: LFHC diet

INTERVENTIONS:
Dietary Supplement: LCHF diet — low-carbohydrate, high-fat (LCHF)diet
Dietary Supplement: LFHC diet — low-fat, high-carbohydrate (LFHC) diet

SUMMARY:
Background:

Researchers want to learn how different diets affect hormone levels, body weight, energy expenditure, liver fat, and more. To do this, they will use specialized techniques and food plans. This is not a weight loss study.

Objective:

To better understand how low-fat and low-carbohydrate foods affect health.

Eligibility:

Men and women ages 18-50 who have a stable body weight and can exercise daily

Design:

Participants will have a screening visit that lasts 4-6 hours. It will include:

Medical history

Physical exam

Fasting blood and urine tests

Questionnaires

Trying foods from the study

Participants will be admitted to the Clinical Center and will stay for 4 weeks without leaving. They can have visitors.

Participants will wear activity and glucose monitors throughout the study. They will be weighed daily and will complete daily exercise. They will eat 3 meals daily, plus snacks. They will give urine, saliva, and blood samples. They will fill out questionnaires and rate their hunger, appetite, and sense of taste. They will have body scans. For the scans, they will lie in a machine that takes X-ray pictures of the body.

Participants will complete activities to measure how many calories they burn and how the diets affect them:

Participants will drink special liquids to measure calories burned, sugar, and sense of taste.

Participants will wear a plastic hood while resting.

Participants will stay alone in a special room for 24 hours.

Participants will eat a low-carb, high-fat diet for 2 weeks and a high-carb, low-fat diet for 2 weeks.

Participants may be dismissed if they purposefully use the study to try to change their body weight.

Sponsoring Institution: National Institute of Diabetes and Digestive and Kidney Diseases

...

DETAILED DESCRIPTION:
Competing theories about obesity and its treatment contrast the relative roles of dietary fat versus carbohydrate on promotion of excessive calorie intake. Advocates of low-carbohydrate diets propose that diets high in carbohydrates lead to elevated insulin secretion and increased calorie intake. Alternatively, proponents of low-fat diets argue that diets high in fat promote passive overconsumption due to the high energy density and low satiety index of high-fat foods. Therefore, we will conduct a feeding study in 20 adult men and women to investigate the differences in ad libitum energy intake resulting from consuming two test diets for a pair of 2-week periods in a randomized, crossover design during a single 4-week inpatient period. The test diets presented to participants will be matched for calories and protein, but the low-carbohydrate diet (approximately10% of calories) will be high in fat (approximately75% of calories) whereas the low-fat diet will be high in carbohydrates (approximately75% of calories) and low in fat (approximately 10% of calories).

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Adults age 18-50 years, male and female
  2. Weight stable (less than or equal to 5 % over past 6 months) as determined by volunteer report
  3. Body mass index (BMI) greater that or equal to 20kg/m2
  4. Body weight greater than or equal to 53 kg
  5. Able to complete daily bouts of stationary cycling at a moderate rate and intensity with a heart rate (HR) equal to or greater than 0.3(SqrRoot) (220-age-HRrest)+HRrest but not exceeding 0.4(SqrRoot) (220-age-HRrest)+HRrest and no signs of arrhythmia

EXCLUSION CRITERIA:

1. Evidence of metabolic or cardiovascular disease, or disease that may influence metabolism (e.g. cancer, diabetes, thyroid disease)
2. Taking any prescription medication or other drug that may influence metabolism (e.g. diet/weight-loss medication, asthma medication, blood pressure medication, psychiatric medications, corticosteroids, or other medications at the discretion of the PI and/or study team)
3. Positive pregnancy test or lactation as determined by volunteer report (women only)
4. Participating in a regular exercise program (> 2h/week of vigorous activity) as determined by volunteer report
5. Hematocrit <37% (women only)
6. Hematocrit < 40% (men only)
7. Caffeine consumption > 300 mg/day as determined by volunteer report
8. Regular use of alcohol (> 2 drinks per day), tobacco (smoking or chewing) amphetamines, cocaine, heroin, or marijuana over past 6 months as determined by volunteer report
9. Psychological conditions such as (but not limited to) eating disorders, claustrophobia, clinical depression, bipolar disorders, that would be incompatible with safe and successful participation in this study, as determined by investigators.

   1. Past or present history of eating disorders as determined by volunteer report
   2. Past or present history of claustrophobia since part of the protocol will involve being confined to a small room for whole-body indirect calorimetry and being in an MRI scanner for liver fat measures
10. Implants, devices, or foreign objects implanted in the body that interfere with the Magnetic Resonance procedures
11. Volunteers with strict dietary concerns (e.g. vegetarian or kosher diet, food allergies)
12. Volunteers unwilling or unable to give informed consent
13. Non-English speakers due to unavailability of required questionnaires in other languages

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hall, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Jaime-Lara RB, Franks AT, Nawal N, Steck MC, Chao AM, Allen C, Brooks BE, Atkinson M, Courville AB, Guo J, Yang S, Marzouk M, Darcey VL, Chung S, Forde CG, Hall KD, Joseph PV. The Role of Diet and Hormones on Taste: Low Carb Compared With Low Fat Study Findings. Curr Dev Nutr. 2025 May 19;9(6):107467. doi: 10.1016/j.cdnut.2025.107467. eCollection 2025 Jun. PMID 40606290
- [Derived] Hengist A, Ong JA, McNeel K, Guo J, Hall KD. Imprecision nutrition? Intraindividual variability of glucose responses to duplicate presented meals in adults without diabetes. Am J Clin Nutr. 2025 Jan;121(1):74-82. doi: 10.1016/j.ajcnut.2024.10.007. Epub 2024 Dec 2. PMID 39755436
- [Derived] Sciarrillo CM, Guo J, Hengist A, Darcey VL, Hall KD. Diet order significantly affects energy balance for diets varying in macronutrients but not ultraprocessing in crossover studies without a washout period. Am J Clin Nutr. 2024 Oct;120(4):953-963. doi: 10.1016/j.ajcnut.2024.08.013. Epub 2024 Aug 18. PMID 39163976
- [Derived] Link VM, Subramanian P, Cheung F, Han KL, Stacy A, Chi L, Sellers BA, Koroleva G, Courville AB, Mistry S, Burns A, Apps R, Hall KD, Belkaid Y. Differential peripheral immune signatures elicited by vegan versus ketogenic diets in humans. Nat Med. 2024 Feb;30(2):560-572. doi: 10.1038/s41591-023-02761-2. Epub 2024 Jan 30. Erratum In: Nat Med. 2024 Jun;30(6):1785. doi: 10.1038/s41591-024-02884-0. PMID 38291301
- [Derived] Sciarrillo CM, Guo J, Hengist A, Darcey VL, Hall KD. Diet order affects energy balance in randomized crossover feeding studies that vary in macronutrients but not ultra-processing. medRxiv [Preprint]. 2023 Oct 4:2023.10.03.23296501. doi: 10.1101/2023.10.03.23296501. PMID 37986904
- [Derived] O'Connor LE, Hall KD, Herrick KA, Reedy J, Chung ST, Stagliano M, Courville AB, Sinha R, Freedman ND, Hong HG, Albert PS, Loftfield E. Metabolomic Profiling of an Ultraprocessed Dietary Pattern in a Domiciled Randomized Controlled Crossover Feeding Trial. J Nutr. 2023 Aug;153(8):2181-2192. doi: 10.1016/j.tjnut.2023.06.003. Epub 2023 Jun 3. PMID 37276937
- [Derived] Hall KD, Guo J, Courville AB, Boring J, Brychta R, Chen KY, Darcey V, Forde CG, Gharib AM, Gallagher I, Howard R, Joseph PV, Milley L, Ouwerkerk R, Raisinger K, Rozga I, Schick A, Stagliano M, Torres S, Walter M, Walter P, Yang S, Chung ST. Effect of a plant-based, low-fat diet versus an animal-based, ketogenic diet on ad libitum energy intake. Nat Med. 2021 Feb;27(2):344-353. doi: 10.1038/s41591-020-01209-1. Epub 2021 Jan 21. PMID 33479499
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-DK-0067.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LCHF Diet Then LFHC Diet | LFHC Diet Then LCHF Diet
Started | 11 | 10
Completed First Phase | 10 | 10
Completed | 10 | 10
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCHF Diet Then LFHC Diet | LFHC Diet Then LCHF Diet | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.7 (7.1) | 31.6 (5.5) | 30.1 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Ad Libitum Energy Intake
Description: Ad libitum energy intake averaged over 14 days for each diet, measured in kilocalories (kcal) per day.
Time Frame: 14 days
Measure: Mean (Standard Error); unit: kcal per day
Groups:
- LC Diet: Low carbohydrate diet
- LF Diet: Low fat diet
Arm/Group | LC Diet | LF Diet
Number analyzed (Participants) | 20 | 20
kcal per day | 2752 (52.0) | 2063 (52.0)

2. Secondary Outcome: Mean Glucose During Oral Glucose Tolerance Test (OGTT)
Description: An OGTT was performed at the end of each 14 day period and the mean glucose was calculated
Time Frame: Day 14
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | LC Diet | LF Diet
Number analyzed (Participants) | 20 | 20
mg/dl | 115.6 (2.9) | 143.3 (2.9)

3. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline to day 14 for each diet, measured in kilograms (kg)
Time Frame: Baseline and day 14
Measure: Mean (Standard Error); unit: kg
Arm/Group | LC Diet | LF Diet
Number analyzed (Participants) | 20 | 20
kg | 1.77 (0.32) | 1.09 (0.32)

4. Secondary Outcome: Change in Body Fat Mass
Description: Change in body fat mass from baseline to day 14 for each diet, measured in kilograms (kg). Body fat mass was measured using Dual-energy X-ray absorptiometry (DXA) measurements.
Time Frame: Baseline and day 14
Measure: Mean (Standard Error); unit: kg
Arm/Group | LC Diet | LF Diet
Number analyzed (Participants) | 20 | 20
kg | -0.18 (0.19) | -0.67 (0.19)

5. Secondary Outcome: Change in Cholesterol
Description: Change in cholesterol from baseline to day 14 for each diet
Time Frame: Baseline and day 14
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | LC Diet | LF Diet
Number analyzed (Participants) | 20 | 20
mg/dl | -1.25 (5.47) | -41.75 (5.47)

6. Secondary Outcome: Change in Triglycerides
Description: Change in triglycerides from baseline to day 14 for each diet
Time Frame: Baseline and day 14
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | LC Diet | LF Diet
Number analyzed (Participants) | 20 | 20
mg/dl | -12.1 (6.4) | 17.9 (6.4)

7. Secondary Outcome: Change in TSH
Description: Change in thyroid stimulating hormone (TSH) from baseline to day 14 for each diet
Time Frame: Baseline and day 14
Measure: Mean (Standard Error); unit: uIU/ml
Arm/Group | LC Diet | LF Diet
Number analyzed (Participants) | 20 | 20
uIU/ml | 0.082 (0.176) | -0.403 (0.176)

8. Secondary Outcome: Change in C-peptide
Description: Change in C-peptide from baseline to day 14 for each diet
Time Frame: Baseline and day 14
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | LC Diet | LF Diet
Number analyzed (Participants) | 20 | 20
ng/ml | -0.610 (0.080) | -0.250 (0.080)

9. Secondary Outcome: Change in CRP
Description: Change in C-reactive protein (CRP) from baseline to day 14 for each diet
Time Frame: Baseline and day 14
Measure: Mean (Standard Error); unit: mg/l
Arm/Group | LC Diet | LF Diet
Number analyzed (Participants) | 16 | 15
mg/l | 0.068 (0.289) | -0.842 (0.296)

ADVERSE EVENTS:
Time Frame: During each 14 day diet period
Arm/Group | LC Diet | LF Diet
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 1/21 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LC Diet (N=21) | LF Diet (N=20)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT03878108/Prot_SAP_000.pdf